CLINICAL TRIAL: NCT01062412
Title: A Single Center, Prospective Clinical Trial to Evaluate the Feasibility of Laser Treatment of the Crystalline Lens to Correct Presbyopia: Philippines
Brief Title: Feasibility Study of Laser Treatment of the Crystalline Lens to Correct Presbyopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No improvement in near vision was detected
Sponsor: LensAR Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52-00013-000 Rev C
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Presbyopia; Cataract
Keywords: Accommodation; Presbyopia; Crystalline lens
MeSH Terms: conditions — Presbyopia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LensAR Laser System — Laser treatment of the crystalline lens

SUMMARY:
The study will evaluate whether the LensAR laser system can be used in the lens of the eye to increase the ability to read and/or see near objects

DETAILED DESCRIPTION:
The objective of this study is to evaluate the feasibility of the LensAR Laser System to surgically intervene within the crystalline lens to improve vision by increasing amplitude of accommodation in patients having elected to undergo lens extraction and IOL implantation

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign and be given a copy of the written informed consent form.
* Subjects must have elected to undergo lens extraction and IOL implantation to treat their ocular disorder then elect to have the LensAR laser surgery as part of the procedure.
* Cataract should not exceed LOCS III Grade 2.
* Subjects must have best corrected distance visual acuity of 20/40 or better in the eye to be treated .
* Subjects must be ≥ 45 years and ≤ 60 years of age at time of subject eligibility visit.
* Subjects must be willing and able to return for scheduled follow up examinations for 6 months after cataract surgery or up to 3 years (at 6 month intervals) if no cataract surgery is performed.
* Subject must have central 7 mm of clear cornea without vascularization

Exclusion Criteria:

* Subjects who are pregnant, lactating, or planning to become pregnant during the course of the study.
* Subjects who have undergone previous corneal or intraocular surgery in the eye to be treated.
* Subjects with a history, signs or symptoms of ocular disease or atypical finding which would be contraindicated under standard of care for cataract surgery.
* Diabetic or hypertensive subjects with clinical evidence of retinal pathology.
* Subjects with macular degenerative pathology.
* Subjects with a history of steroid-responsive rise in IOP or uncontrolled glaucoma in either eye.
* Subjects with known lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Subjects with corneal disease or pathology that precludes applanation of the cornea or transmission of laser wavelength or distortion of laser light.
* Subjects who cannot attain ocular dilation adequate to allow laser treatment within the minimum range based on the laser procedure to be applied.
* Subjects with known sensitivity to planned study concomitant medications.
* Subjects using systemic medication that is known to reduce the amplitude of accommodation (such as medication for motion sickness containing hyoscine or other antimuscarinic drugs, anticholinergic drugs, anti-psychotic drugs, tricyclic antidepressants and other drugs acting on the central nervous system).
* Subjects participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10-04 (Actual); Study Completion 2011-10-04 (Actual)

PRIMARY OUTCOMES:
Increased objective amplitude of accommodation | 1 month

SECONDARY OUTCOMES:
Rate of adverse events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Uy, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines